CLINICAL TRIAL: NCT03795025
Title: ContraTRAIN - a Validation Study of Contralateral Training Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Trainome 2019#014
Record Dates: First submitted 2018-12-21; First posted 2019-01-07 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Contralateral; Strength training; Muscle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3x10RM + no training (Experimental)
  Interventions: Other: Strength training 3x10RM + no training
- 6x10RM + no training (Experimental)
  Interventions: Other: Strength training 6x10RM + no training
- 3x10RM + 6x10RM (Experimental)
  Interventions: Other: 3x10RM + 6x10RM
- Control (No Intervention): This arm includes 3 weeks of testing and 7 weeks of no intervention and post tests, followed by 7 weeks of progressive unilateral strength training 3 times per week for 7 weeks. Both legs exercises individually with 3 sets of 10 maximal repetitions.

INTERVENTIONS:
Other: Strength training 3x10RM + no training — Progressive unilateral strength training 3 times per week for 3 + 7 weeks. One leg exercises with 3 sets of 10 maximal repetitions, the other leg does not exercise.
  Arms: 3x10RM + no training
Other: Strength training 6x10RM + no training — Progressive unilateral strength training 3 times per week for 3 + 7 weeks. One leg exercises with 6 sets of 10 maximal repetitions, the other leg does not exercise.
  Arms: 6x10RM + no training
Other: 3x10RM + 6x10RM — Progressive unilateral strength training 3 times per week for 3 + 7 weeks. One leg exercises with 3 sets of 10 maximal repetitions, the other leg exercises with 6 sets of 10 maximal repetitions.
  Arms: 3x10RM + 6x10RM

SUMMARY:
This study aims to validate the use of contralateral designs in studies of effects of resistance exercise. It will recruit healthy young (18-35 years) individuals, which will be allocated to 4 experimental groups. In two of the experimental groups, 3x10 or 6x10 repetitions of heavy resistance exercise on one leg will be combined with no training of the other leg for 7 weeks. In the third group, 3x10 repetitions of heavy resistance exercise on one leg will be combined with 6x10 repetitions of heavy resistance exercise on the other leg for 7 weeks. In the fourth group, which serves as a control group, a period of no training (similar in length to the training period of groups 1-3; 7 weeks), before both legs will train 3x10 repetitions of heavy resistance exercise in an unilateral manner.

DETAILED DESCRIPTION:
Our understanding of how exercise affects muscular adaptations at the cellular and molecular level comes from the use of skeletal muscle biopsies. Such studies are met by several challenges, including its invasive nature, costs of muscle analyses, large inter-participant variability in response to exercise and a limited number of subjects (related to ethical concerns regarding exposing participants to biopsies). Consequently, studies often include small sample sizes, resulting in low statistical power. This poses a great challenge to the field of exercise physiology. While increasing sample size may not always be feasible, employing alternative designs may offer a way to increase the statistical power. An example of such a design is the so-called cross-over design, wherein participants serve as their own control thereby reducing the inter-participant variation. An interesting variant of the cross-over design is the unilateral or contralateral exercise model. In such designs, each of the participant's limbs (e.g. legs) are randomly allocated to perform different types of training/treatments in close temporal proximity. This design obliterates the need for a wash-out period and removes the potential effects of confounding factors such as diet, activity and sleep decreases. Thus, resources, time spent and variability can be reduced. However, validation of such studies is lacking.

In an effort to validate a contralateral training design, the investigators will recruit young (18-35 years) healthy individuals to 4 groups performing unilateral progressive strength training; (1) one leg with no training and one leg with 3x10 maximal repetitions, (2) one leg with no training and one leg with 6x10 maximal repetitions, (3) one leg with 3x10 maximal repetitions and one leg with 6x10 maximal repetitions and (4) a control group with an initial period of no training (similar in length to the training period of groups 1-3) followed by a period of 3x10 maximal repetitions on each leg. Leg training will consist of one-legged leg press and one-legged knee extensions. All groups, except the control group (during the no-training control period), will train the upper body by 3x10 maximal repetitions in bench press and lying rowing. Prior to the 7 week training intervention, all four groups will go through a 3-week period of familiarization to training and repeated testing (4 test time points for performance measures).

This design allows us to investigate the benefits of a contralateral design compared to the more common two-group design, the intra-individual variation vs the inter-individual variation, the potential contralateral effect of training one leg on the physiology and functional abilities of the non-trained leg, and whether or not these perspective are affected by training volume. We will also investigate whether participant classification into low or high responders is universal across several measures of muscle mass and strength, and between different training volumes. Further, by measuring several hypertrophy-related outcomes (e.g. changes in ribosome volume, activation of satellite cells and transcriptional changes), the investigators will extend previous findings regarding the effects of training volume on these variables and their ability to predict training outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Smoking
* Strength training more than 2 times per months for the last 6 months
* Endurance training more than 3 hours per week
* Adverse reactions to lidocaine
* Consumption of supplements or medication affecting muscular adaptations to strength training

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Muscle fiber area | Changes over the course of the intervention (0-10 weeks)
  Muscle cell cross-sectional area measured in biopsies from m. vastus lateralis using immunohistochemistry

SECONDARY OUTCOMES:
Body mass composition | Changes over the course of the intervention (0-10 weeks)
  Body mass composition measured using Dual-energy X-ray absorptiometry (DXA)
Rate of muscle protein synthesis (%/day) | Mesured over 3 days in week 7 of the study
  By ingesting deuterium we will label alanine to measure the rate of its incorporation into muscle proteins. This is done by collection of blood before, during and after, and a biopsy 3 days after deuterium ingestion to be analyzed with chromatography and mass spectrometry. Results will be reported as a rate of synthesis in %/day.
M. vastus lateralis thickness | Changes over the course of the intervention (0-10 weeks)
  M. vastus lateralis thickness mesured by ultrasound
Unilateral leg press strength (1RM test) | Changes over the course of the intervention (0-10 weeks)
  The ability of muscles of the lower body to exert maximal force during dynamic movements in a leg press
Unilateral knee extension strength (1RM test) | Changes over the course of the intervention (0-10 weeks)
  The ability of muscles of the lower body to exert maximal force during dynamic movements in a knee extension
Barbell bench press muscle strength (1RM test) | Changes over the course of the intervention (0-10 weeks)
  The ability of muscles of the upper body to exert maximal force during dynamic movements in a bench press
Lying rowing muscle strength (1RM test) | Changes over the course of the intervention (0-10 weeks)
  The ability of muscles of the upper body to exert maximal force during dynamic movements in a lying row exercise
Unilateral lower body isokinetic muscle strength at 60 and 240 deg per second in a mechanical dynamometer (Humac NORM) | Changes over the course of the intervention (0-10 weeks)
  The ability of muscles of the lower body to exert maximal force during isokinetic movements
Unilateral lower body isometric muscle strength in a mechanical dynamometer (Humac NORM) | Changes over the course of the intervention (0-10 weeks)
  The ability of muscles of the lower body to exert maximal force during isometric contractions
One-legged cycling | Changes over the course of the intervention (0-10 weeks)
  Performance indicies measured during an incremental one-legged cycling test
Muscle phenotype | Changes over the course of the intervention (0-10 weeks)
  Muscle fiber type composition measured in biopsies from m. vastus lateralis using immunohistochemistry
Muscle cell biological traits | Changes over the course of the intervention (0-10 weeks)
  Muscle cell biological traits, including numbers of myonuclei, satelitte cells and capillaries, measured in biopsies from m. vastus lateralis using immunohistochemistry
Gene expression in skeletal muscle | Changes over the course of the intervention (0-10 weeks)
  RNA (e.g. messenger RNA, ribosomal RNA, microRNA, long non-coding RNA) abundances in m. vastus lateralis, measured both as single genes and at the level of the transcriptome
Protein abundances in skeletal muscle measured by western blot | Changes over the course of the intervention (0-10 weeks)
  Levels of proteins and their modification status (e.g. phosphorylation) in m. vastus lateralis, measured at the level of single proteins and at the level of the proteome
Hormones in blood | Changes over the course of the intervention (0-10 weeks)
  Levels of hormones in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to the academic community through the general biobank "The Trainsome - effects of exercise and environment on human cells" (REK-2013/2045, Regional Comitees for Medical and Health Research Ethics South East). Data will be available on request and will be restricted to scientists and/or projects with a sound scientific purpose and rationale.